CLINICAL TRIAL: NCT04519502
Title: Maternal Morbidity and Mortality During the COVID-19 Pandemic
Acronym: MFMU COVID-19
Status: Completed | Type: Observational
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: HD36801 - MFMU COVID-19; U01HD036801 (NIH)
Record Dates: First submitted 2020-08-18; First posted 2020-08-19 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; Pregnancy Complications
MeSH Terms: conditions — COVID-19; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Randomly Selected Delivery Dates 2019: Women who deliver at one of the MFMU Network hospitals on randomly selected days between March 1 and December 31, 2019.
- Randomly Selected Delivery Dates 2020: Women who deliver at one of the MFMU Network hospitals on randomly selected days between March 1 and December 31, 2020
- Confirmed COVID-19 Infections: Women with confirmed COVID-19 infection between March 1, 2020 and December 31, 2020 and who delivered on or before December 31, 2020.

SUMMARY:
A cohort study of women who deliver at select sites on randomly selected days in 2019 and 2020, and all confirmed COVID-19 infections among pregnant or immediately postpartum women in 2020. The study population includes approximately 24,400 deliveries on randomly selected days in 2019 and 2020, and an additional 1000-2100 confirmed COVID-19 infections among pregnant women or immediately postpartum.

DETAILED DESCRIPTION:
This cohort study includes women who deliver at one of the MFMU Network hospitals on randomly selected days between March 1 and December 31, 2019 and March 1 and December 31, 2020 to evaluate the effect of a major public health crisis (COVID-19 pandemic) on maternal morbidity and mortality among pregnant and immediately postpartum women. This time period allows for calendar months in 2020 representing the key time period of the pandemic - after testing became available and changes were implemented in healthcare. Inclusion of the same months from 2019 represent the time period prior to the pandemic.

In addition to the cohort of women delivering at the selected MFMU Network sites on randomly selected days, all pregnant and immediately postpartum (within 6 weeks of delivery) with confirmed COVID-19 infection will be included in this study. Both women who were managed in-patient and those managed out-patient with COVID-19 infection will be included. All pregnant women with confirmed COVID-19 infection between March 1, 2020 and December 31, 2020 will be followed for maternal and neonatal outcomes through 6 weeks after delivery or surgical removal of the pregnancy.

Trained research staff will abstract data from the hospital's electronic medical records that meet eligibility criteria. Measures of healthcare and community-based modifications in response to the pandemic will be recorded by research staff. Individual participant data will include baseline data, COVID-19 exposure data, and maternal and neonatal outcome data.

The three primary objectives are 1) to evaluate whether pregnant or immediately postpartum women experience higher maternal morbidity and mortality during the COVID-19 pandemic than before the pandemic, 2) to evaluate whether women with COVID-19 infection, both in- and out-patient, have higher maternal morbidity and mortality than pregnant women without COVID-19 infection, and 3) to describe maternal and neonatal outcome data for all pregnant and immediately postpartum women with a confirmed COVID infection and contribute these data to an NICHD COVID-19 pregnancy registry. The primary endpoint, maternal morbidity and mortality, is defined as morbidity related to hypertensive disorders of pregnancy, morbidity related to postpartum hemorrhage, or morbidity related to infection during pregnancy or within six weeks (42 days) postpartum. For primary objective 1, the study has more than 90% power to show a 30% increase in the rate of the primary endpoint assuming the rate is at least 3% in calendar year 2019 and an alpha of 0.05 two-sided. For primary objective 2, the study will have more than 85% power to detect a 50% increase in the primary composite maternal morbidity endpoint, from 5% to 7.5% with an alpha=0.05 two sided if only 1,000 confirmed COVID-19 people are enrolled (80% power to detect a 30% increase in the primary composite if 2,200 confirmed COVID-19 people are enrolled).

For objective 1, analyses of the primary endpoint will consist of summarizing the proportions of participants with the primary endpoint for each calendar year cohort and calculating the corresponding relative risks with 95% confidence intervals. Individual morbidity composites (hypertensive disorders, postpartum hemorrhage, and infection) will also be compared by calendar year cohort. Outcome rates within 2019 will be graphically displayed and tested over time to ensure changes are not evident during the year that may explain differences between calendar years 2019 and 2020. For objective 2, analyses of the primary endpoint will consist of summarizing the proportions of participants with the primary endpoint among women with confirmed COVID-19 infection and those without confirmed infection, and calculating the corresponding relative risk with 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Women who deliver at a selected hospital participating in the MFMU Network on selected dates sent by the Data Coordinating Center from March 1, 2019, through Dec, 31, 2019. Women delivered in the calendar year 2019 will serve as the controls (before pandemic).
* Women who deliver at a selected hospital participating in the MFMU Network on selected dates sent by the Data Coordinating Center from March 1, 2020, through Dec, 31, 2020. Women delivered in the calendar year 2020 will be considered as deliveries during the pandemic (research question 1) and non-confirmed positives as controls (research question 2).
* Pregnant and postpartum (within 6 weeks of delivery) women with confirmed COVID-19 infection from March 1, 2020, through Dec, 31, 2020 and who deliver on or before December 31, 2020. Both those with COVID-19 infection requiring in-patient management and those managed as out-patients will be included. Confirmed COVID-19 infection is defined as a positive COVID-19 viral (i.e., nucleic acid or antigen tests) test during pregnancy through 42 days postpartum.

Exclusion Criteria:

* Multifetal gestation higher than twins

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 24,400 deliveries on randomly selected days in 2019 and 2020, and an additional 1000-2100 confirmed COVID-19 infections among pregnant women or immediately postpartum
Sampling Method: Probability Sample
Enrollment: 25604 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
Maternal Mortality and Morbidity Composite | During pregnancy through 6 weeks postpartum
  Percentage of patients with at least one of the following: mortality, morbidity related to hypertensive disorders of pregnancy, morbidity related to postpartum hemorrhage, morbidity related to infection

SECONDARY OUTCOMES:
Cesarean Delivery | Delivery
  Percentage of patients that had cesarean delivery
Severe maternal morbidity or mortality | During pregnancy through 6 weeks postpartum
  Percentage of patients with at least one of teh following: death, ICU admission, transfusion of 4 or more units of packed red blood cells
Adverse maternal outcomes | During pregnancy through 6 weeks postpartum
  a. Percentage of patients with the following outcomes: ICU admission, ventilator support, extracorporeal membrane oxygenation (ECMO), pressor support, cardiomyopathy, venous thromboembolism (deep venous thrombosis or pulmonary embolus), arterial thrombosis including cerebrovascular accident, cerebral venous sinus thrombosis, renal failure requiring dialysis, encephalopathy, superficial or deep incisional surgical site infection, multisystem inflammatory syndrome
Adverse neonatal outcomes | Delivery through hospital discharge up to 120 days
  a. Percentage of neonates with the following outcomes: fetal or neonatal death, preterm birth < 37 weeks gestation, small for gestational age, major congenital malformations, perinatal preterm composite (defined as fetal or neonatal death, severe bronchopulmonary dysplasia, intraventricular hemorrhage grades III-IV, necrotizing enterocolitis, periventricular leukomalacia, retinopathy of prematurity stage III-V, or proven sepsis), perinatal term composite (defined as fetal or neonatal death, respiratory support within first 72 hours, Apgar score <=3 at 5 minutes, hypoxic ischemic encephalopathy, seizure, infection, birth trauma, meconium aspiration syndrome, intracranial or subgaleal hemorrhage, or hypotension requiring vasopressor support
Neonatal infection | Delivery through hospital discharge up to 120 days
  Percentage of neonates with infection diagnosed within delivery hospitalization
Maternal in-patient hospitalization days | During pregnancy through 6 weeks postpartum
  Number of maternal in-patient hospitalization days
Maternal ICU admission | During pregnancy through 6 weeks postpartum
  Percentage of patients admitted to the ICU
Duration of labor and delivery | During pregnancy through delivery
  Length of time on labor and delivery from admission to delivery for the delivery hospitalization
Neonatal length of stay | Delivery through hospital discharge up to 120 days
  Length of time from delivery to hospital discharge
Neonatal ICU length of stay | Delivery through hospital discharge up to 120 days
  Length of time from neonatal ICU admission to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Monica Longo, MD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Torri Metz, MD, Study Chair — University of Utah Medical Center
Locations (12):
- United States (12):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois
  - Columbia University-St. Luke's Hospital, New York, New York
  - University of North Carolina-Chapel Hill, Chapel Hill, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - Brown Univeristy, Providence, Rhode Island
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared per NIH policy.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Metz TD, Clifton RG, Hughes BL, Sandoval GJ, Grobman WA, Saade GR, Manuck TA, Longo M, Sowles A, Clark K, Simhan HN, Rouse DJ, Mendez-Figueroa H, Gyamfi-Bannerman C, Bailit JL, Costantine MM, Sehdev HM, Tita ATN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Association Between Giving Birth During the Early Coronavirus Disease 2019 (COVID-19) Pandemic and Serious Maternal Morbidity. Obstet Gynecol. 2023 Jan 1;141(1):109-118. doi: 10.1097/AOG.0000000000004982. Epub 2022 Oct 27. PMID 36357949